CLINICAL TRIAL: NCT00154947
Title: Develop Biomarkers for Assessing RA Joint Erosion
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Palo Alto Medical Foundation (Other)
Other Study IDs: 9361700330
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-07-20 (Estimated); Status verified 2006-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
With the current therapeutic focus in rheumatoid arthritis (RA) shifting from symptom control to actual disease modification there is a growing demand for more objective and sensitive ways to evaluate structural damage in the joints of these RA patients. Conventional radiography of bone erosion and joint-space narrowing was the only imaging approach available for this. Now significant advantages are offered in terms of speed, precision and scope over conventional methods. These advances include digital radiography and computer aided analysis as well as MRI which allow earlier identification of bone erosion and direct visualization of pre-erosive changes, such as bone inflammation and synovitis. Molecular markers of tissue turnover have been used for decades in clinical trials of osteoporosis, but only recently in RA. In contrast to serum C-reactive protein (CRP), which is only a nonspecific indicator of systemic inflammation and not directly reflective of structural damage to joints, more recently developed molecular markers of synovial, cartilage and bone turnover might provide a better indication of destructive activity of the disease. Compared with radiography and MRI assessment, molecular markers are particularly useful for patient selection and treatment, but can be used in a variety of ways to accelerate clinical trials and reduce the uncertainty and cost of drug development. In this project, we will set up a panel of molecular markers which could show an association with the MRI results and have a quantitative correlation with the degree of joint damage (sensitivity: 90 - 95%; specificity: 80 - 90%). The work in this project includes imaging markers evaluation and molecular markers analysis: X-ray scoring; MRI; Bone degradation markers; Bone formation; Cartilage degradation; Cartilage synthesis; Synovial turnover and Others. Nine molecular markers will be examined: CartiLaps ELISA/CTX-II, Urinary CrossLaps ELISA/CTX-I, and Serum osteocalcin, Serum COMP, MMP-3, Serum PINP, Serum PICP, Urinary PIIINP and Serum YKL-40. The data will be managed to evaluate the significance of correlation to image and clinical reports, so as to get a simple algorithm of parameters (molecular markers) which can reflect the structural damage of joint using mathematics and computer science.

DETAILED DESCRIPTION:
With the current therapeutic focus in rheumatoid arthritis (RA) shifting from symptom control to actual disease modification there is a growing demand for more objective and sensitive ways to evaluate structural damage in the joints of these RA patients. Conventional radiography of bone erosion and joint-space narrowing was the only imaging approach available for this. Now significant advantages are offered in terms of speed, precision and scope over conventional methods. These advances include digital radiography and computer aided analysis as well as MRI which allow earlier identification of bone erosion and direct visualization of pre-erosive changes, such as bone inflammation and synovitis. Molecular markers of tissue turnover have been used for decades in clinical trials of osteoporosis, but only recently in RA. In contrast to serum C-reactive protein (CRP), which is only a nonspecific indicator of systemic inflammation and not directly reflective of structural damage to joints, more recently developed molecular markers of synovial, cartilage and bone turnover might provide a better indication of destructive activity of the disease. Compared with radiography and MRI assessment, molecular markers are particularly useful for patient selection and treatment, but can be used in a variety of ways to accelerate clinical trials and reduce the uncertainty and cost of drug development. In this project, we will set up a panel of molecular markers which could show an association with the MRI results and have a quantitative correlation with the degree of joint damage (sensitivity: 90 - 95%; specificity: 80 - 90%). The work in this project includes imaging markers evaluation and molecular markers analysis: X-ray scoring (bone erosion and joint-space narrowing); MRI (bone erosion, synovitis, cartilage erosion, tendonitis, ligament rupture); Bone degradation markers (CTX-I, NTX-I, DPD); Bone formation (osteocalcin, alkaline phosphatase, PICP, PINP); Cartilage degradation (CTX-II, COMP); Cartilage synthesis (PIICP, PIINP, glycosaminoglycan); Synovial turnover (Glc-Gal-PYD) and Others (Hyaluronic acid, YKL-40, MMP-1, MMP-3, MMP-13, TIMPs and type III collagen N-propeptide). Nine molecular markers (including bone formation and degradation, cartilage synthesis and degradation) will be examined: CartiLaps ELISA/CTX-II, Urinary CrossLaps ELISA/CTX-I, and Serum osteocalcin, Serum COMP, MMP-3, Serum PINP, Serum PICP, Urinary PIIINP and Serum YKL-40. The data will be managed to evaluate the significance of correlation to image and clinical reports, so as to get a simple algorithm of parameters (molecular markers) which can reflect the structural damage of joint using mathematics and computer science.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis

Exclusion Criteria:

* Nil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-05; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Liang-In Lin, PhD, Principal Investigator — Department of Clinical Laboratory Sciences and Medical Biotechnology, National Taiwan University
Locations (1):
- Liang-In Lin, Taipei, Taiwan